CLINICAL TRIAL: NCT02281019
Title: Clinical Registry of Cholangioscopy Using the SpyGlass™ Direct Visualization System (DVS) Throughout the AMEA (Asia, Middle-East, Africa) Region
Brief Title: SpyGlass AMEA Registry
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90947376
Record Dates: First submitted 2014-10-09; First posted 2014-11-03 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Biliary Stricture; Biliary Obstruction Due to Common Bile Duct Stone; Periampullary Tumor; Hemobilia
MeSH Terms: conditions — Hemobilia | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Tissue acquisition in the bile ducts
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Indeterminate strictures or undefined filling defects
  Interventions: Procedure: ERCP (Endoscopic Retrograde Cholangiopancreatography); Device: SpyGlass DVS and SpyGlass Digital Simple (DS)
- Biliary stone cases
  Interventions: Procedure: ERCP (Endoscopic Retrograde Cholangiopancreatography); Device: SpyGlass DVS and SpyGlass Digital Simple (DS)
- Other indications
  Interventions: Procedure: ERCP (Endoscopic Retrograde Cholangiopancreatography); Device: SpyGlass DVS and SpyGlass Digital Simple (DS)

INTERVENTIONS:
Procedure: ERCP (Endoscopic Retrograde Cholangiopancreatography) — ERCP procedure will be performed to visualize bile ducts.
Device: SpyGlass DVS and SpyGlass Digital Simple (DS) — Cholangioscopy using SpyGlass™ DVS or SpyGlass DS will be performed post ERCP for direct viewing of the bile ducts. What is seen during the procedure will determine a course of treatment. Among the options are biopsies taken, stones treated/removed, or a stent placed

SUMMARY:
The purpose of this study is to document indications for cholangioscopy and clinical utility of the SpyGlass Direct Visualization System (DVS) throughout the AMEA (Asia, Middle-East, Africa) region when used per standard of practice.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Willing and able to provide written informed consent to participate in the study.
* Willing and able to comply with the study procedures.
* Indicated for ERCP and cholangioscopy or indicated for ERCP with suspected need for cholangioscopy.

Exclusion Criteria:

* Endoscopic techniques are contraindicated.
* ERCP is contraindicated
* A medical condition that warrants the use of the device outside of the indication for use.
* Requirement for anticoagulation that cannot be safely stopped at least 7 days prior to the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients seen at an investigational site during the enrollment period
  * Presenting with an indication for cholangioscopy, or
  * Presenting with a possible indication for cholangioscopy to be determined during the ERCP procedure immediately preceding the SpyGlass procedure.
Sampling Method: Non-Probability Sample
Enrollment: 526 (Actual)
Dates: Start 2014-11-15 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10-18 (Actual)

PRIMARY OUTCOMES:
Procedural success for indeterminate strictures or undefined filling defects | Procedure - the average expected duration of the procedure is 1.5 hours
  For indeterminate strictures or undefined filling defects cases procedural success is defined as 1) ability to visualize stricture or defect, and 2) ability to provide visual impression of malignancy, and 3) when applicable, ability to obtain SpyBite biopsy adequate for histology
Procedural success for biliary stone cases | Procedure - the average expected duration of the procedure is 1.5 hours
  For biliary stone cases procedural success is defined as 1) ability to visualize the stone(s), and 2) ability to successfully initiate stone fragmentation, and 3) ability to achieve stone clearance in one or more SpyGlass procedures.
Procedural success for other indications | Procedure - the average expected duration of the procedure is 1.5 hours
  For other indications procedural success is defined as ability to establish diagnosis and /or complete therapy in the following categories: 1) pre-operative assessment of extent of peri-ampullary and biliary tumors, 2) selective guidewire placement, 3) assessment of unexplained hemobilia, 4) assessment of portal biliopathy, 5) assessment of intraductal biliary ablation therapy, 6) extraction of migrated stents, or 7) other.

SECONDARY OUTCOMES:
Evaluation of serious adverse events (SAEs) related to the SpyGlass devices and/or the SpyGlass procedure | Procedure from enrollment through the 72 Hour Post Procedure Follow-up Visit
  Evaluation of serious adverse events (SAEs) related to the SpyGlass devices and/or the SpyGlass procedure from enrollment through the 72 Hour Post Procedure Follow-up Visit.
Impact of SpyGlass procedure on suspected diagnosis based on prior ERCP | Procedure - the average expected duration of the procedure is 1.5 hours
Evaluation of impact of use of antibiotics on incidence of SAEs related to the device and/or procedure. | Procedure - the average expected duration of the procedure is 1.5 hours
For patients undergoing SpyBite biopsy: correlation between number of biopsies and conclusive histopathology of SpyBite biopsies. | Procedure to 6 months
  Assessment Detail:
  Endpoint determined for all patients in whom SpyBite biopsy was taken and observed image features were reported.
  Observed image features include the following categories: None, Growth, Stricture, Hyperplasia, Ulceration, Mass, Dilated tortuous vessels, Papillary or villous projections, Intraductal nodules, Mucus.
For patients undergoing stone management: number of SpyGlass procedures needed to reach stone clearance. | Procedure - the average expected duration of the procedure is 1.5 hours
For patients undergoing stone management: correlation between stone size and ability to reach stone clearance in one SpyGlass session. | Procedure - the average expected duration of the procedure is 1.5 hours
For patients undergoing stone management: incidence of visualization of stones not suspected during previous ERCP. | Procedure - the average expected duration of the procedure is 1.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Benedict Devereaux, Principal Investigator — Royal Brisbane and Women's Hospital; James Lau, Principal Investigator — Prince of Wales Hospital; Randhir Sud, Principal Investigator — Institute of Digestive & Hepatobiliary Sciences; Saad Niaz, Principal Investigator — Civil Hospital Karachi; Abdulrahman Aljebreen, Principal Investigator — King Khalid University Hospital; Ang Tiing Leong, Principal Investigator — Changi General Hospital Pte Ltd.; Jorg Reichenberger, Principal Investigator — Netcare Unitas Hospital; Jong Moon, Principal Investigator — Soon Chun Hyang University; Rungsun Rerknimitr, Principal Investigator — King Chulalongkorn Memorial Hospital; Ichiro Yasuda, Principal Investigator — Teikyo University Mizonokuchi Hospital; Arthur J. Kaffes, Principal Investigator — Royal Prince Alfred Hospital, Sydney, Australia; Nam Q. Nguyen, Principal Investigator — Royal Adelaide Hospital; Amit Maydeo, Principal Investigator — Baldota Institute of Digestive Sciences; Mohan Ramchandani, Principal Investigator — Asian Institute of Gastroenterology; Mahesh Goenka, Principal Investigator — Apollo Gleneagles Hospital; Professor R. Kochhar, Principal Investigator — Postgraduate Institute of Medical Education & Research; Takao Itoi, Principal Investigator — Tokyo Medical University; Masayuki Kitano, Principal Investigator — Kinki University School of Medicine; Jong K. Lee, Principal Investigator — Samsung Medical Center; Dongwan Seo, Principal Investigator — Asan Medical Center
Locations (20):
- Australia (3):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital, Adelaide
  - Royal Prince Alfred Hospital, Newtown
- Prince of Wales Hospital, Shatin, Hong Kong
- India (5):
  - Apollo Gleneagles Hospitals Kolkata, Kolkata, West Bengal
  - Postgraduate Institute of Medical Education & Research, Chandigarh
  - Medanta -The Medicity Institute of Digestive & Hepatobiliary Sciences, Gūrgaon
  - Asian Institute of Gastroenterology, Hyderabad
  - Baldota Institute of Digestive Sciences, Pārel
- Japan (3):
  - Teikyo University Mizonokuchi Hospital, Kawasaki
  - Kinki University School of Medicine, Ōsaka-sayama
  - Tokyo Medical University, Tokyo
- Civil Hospital- Karachi, Karachi, Pakistan
- King Khalid University Hospital, Riyadh, Saudi Arabia
- Changi General Hospital Pte Ltd., Singapore, Singapore
- Netcare Unitas Hospital, Centurion, South Africa
- South Korea (3):
  - Soon Chun Hyang University Bucheon Hospital, Bucheon-si
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand

REFERENCES:
- [Derived] Maydeo AP, Rerknimitr R, Lau JY, Aljebreen A, Niaz SK, Itoi T, Ang TL, Reichenberger J, Seo DW, Ramchandani MK, Devereaux BM, Lee JK, Goenka MK, Sud R, Nguyen NQ, Kochhar R, Peetermans J, Goswamy PG, Rousseau M, Bhandari SP, Angsuwatcharakon P, Tang RSY, Teoh AYB, Almadi M, Lee YN, Moon JH; SpyGlass AMEA Registry Group. Cholangioscopy-guided lithotripsy for difficult bile duct stone clearance in a single session of ERCP: results from a large multinational registry demonstrate high success rates. Endoscopy. 2019 Oct;51(10):922-929. doi: 10.1055/a-0942-9336. Epub 2019 Jun 27. PMID 31250408